CLINICAL TRIAL: NCT04434105
Title: Ultrasound-guided PRP Versus Steroid Injections in Management of Carpal Tunnel Syndrome; a Comparative Study
Brief Title: Ultrasound-guided PRP Versus Steroid Injections in Management of Carpal Tunnel Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Hassan Abu-Zaid, principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-06-14; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: PRP injection; Local injection; CTS
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Triamcinolone Acetonide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP group (Experimental): patients received ultrasound-guided injection of 2 mL PRP into the affected carpal tunnel.patients will be injected twice with 2 weeks intervals
  Interventions: Drug: platlet rich plasma (PRP)
- Steroid group (Active Comparator): patients received ultrasound-guided injection of 2 mL steroids (40 mg triamcinolone acetonide). into the affected carpal tunnel. patients will be injected twice with 2 weeks intervals
  Interventions: Drug: Triamcinolone Acetonide
- Control group (Placebo Comparator): patients received ultrasound-guided injection of 2 mL saline patients will be injected twice with 2 weeks intervals
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: platlet rich plasma (PRP) — Platelet-rich plasma (PRP) promotes angiogenesis, neurogenesis, and nerve regeneration, also it could reduce swelling and inflammation of the flexor tenosynovitis.
  Arms: PRP group
Drug: Triamcinolone Acetonide — 40 mg triamcinolone acetonide
  Arms: Steroid group
Drug: Saline — Saline
  Arms: Control group

SUMMARY:
Patients will be randomly divided into 3 equal groups: Group I received ultrasound guided injection of 2 mL PRP into the affected carpal tunnel. Group II received ultrasound guided injection of 2 mL steroids (40 mg triamcinolone acetonide). Group III received ultrasound guided injection of 2 mL saline as placebo control.

DETAILED DESCRIPTION:
Patients will be randomly divided into 3 equal groups: Group I received ultrasound guided injection of 2 mL PRP into the affected carpal tunnel. Group II received ultrasound guided injection of 2 mL steroids (40 mg triamcinolone acetonide). Group III received ultrasound guided injection of 2 mL saline as placebo control.

Each group will be injected twice with 2 weeks intervals. All procedures were done after informed consent. Evaluation of the patients at baseline, 3 and 6 months after last injection was done clinically by measuring visual analogue scale (VAS), electrophysiologically (by measuring motor and sensory nerve conduction studies of median nerve using a standardized technique) and ultrasonographic study by measuring cross sectional area (CSA) of median nerve at the level of pisiform.

ELIGIBILITY:
Inclusion Criteria:

* mild or moderate idiopathic CTS (diagnosed clinically, ultrasonography & electrophysiologically and classified according to the American Association of neuromuscular diagnostic medicine monograph).

Exclusion Criteria:

* Patients with severe or secondary type of CTS

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | Change from 3 months after last injection and 6 months after last injection
  Scale for assessement the degree of pain along 0-10 scale
measuring motor and sensory nerve conduction studies of median nerve using a standardized technique | Change from 3 months after last injection and 6 months after last injection
  electrophysiologically by measuring motor and sensory nerve conduction studies of median nerve using a standardized technique
cross-sectional area (CSA) of the median nerve at the level of the pisiform. | Change from 3 months after last injection and 6 months after last injection
  ultrasonographic study by measuring cross-sectional area (CSA) of the median nerve at the level of the pisiform.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malahias MA, Johnson EO, Babis GC, Nikolaou VS. Single injection of platelet-rich plasma as a novel treatment of carpal tunnel syndrome. Neural Regen Res. 2015 Nov;10(11):1856-9. doi: 10.4103/1673-5374.165322. PMID 26807124
- See also: effect of PRP on CTS — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4705801/